CLINICAL TRIAL: NCT04074538
Title: The National Colorectal Cancer Cohort Study-Precision Medical Research in Colorectal Cancer
Brief Title: the National Colorectal Cancer Cohort (NCRCC) Study: National Colorectal Cancer Research Consortium
Status: Recruiting | Type: Observational
Sponsor: Ding Ke-Feng (Other)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); West China Hospital (Other); Sun Yat-sen University (Other); Shanghai Zhongshan Hospital (Other); Peking University People's Hospital (Other); Peking University Cancer Hospital & Institute (Other); Fujian Cancer Hospital (Other Government); Hubei Cancer Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Shanxi Province Cancer Hospital (Other); Changhai Hospital (Other); Zhejiang Cancer Hospital (Other); Third Affiliated Hospital of Third Military Medical University (Other); Air Force Military Medical University, China (Other); Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor-Investigator, Ding Ke-Feng, Professor, Zhejiang University
Organization: Zhejiang University (Other)
Other Study IDs: CRCCZ-ncrcc
Record Dates: First submitted 2019-08-26; First posted 2019-08-30 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; cohort study; CRC screening
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Formalin fixed and paraffin embedded (FFPE) and fresh frozen tissue (multiple sources/locations) from the tumor, blood, urine, feces
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
NCRCC study is a national prospective cohort study including colorectal cancer screening population and stage Ⅰ-Ⅳ colorectal cancer patients.

DETAILED DESCRIPTION:
NCRCC study is a large-scale multicenter study which includes 16 hospitals and research centers, establishing a national cohort which consists of two subcohorts (CRC Screening Cohort and Colorectal Cancer Patient Cohort).

1. To assess risk factors for colorectal cancer and evaluate risk prediction model of colorectal cancer to identify the high-risk population.
2. To discover, test and validate new biological markers (e.g. genetic, epigenetic, transcriptomic, metabolomics, proteomic and metagenomics biomarkers) for early diagnosis, prediction of clinical outcomes (e.g. therapeutic response, toxicity, surgical complications) and survivorship endpoints (e.g. recurrence, survival, quality of life, second primary cancer).
3. To estimate associations of epidemiological determinants (e.g. medication and supplement use, diet, lifestyle pattern) with clinical outcomes and survivorship endpoints among CRC patients.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Mentally/physically able to consent and participate
* Subjects aged ≥18 years old (Colorectal Cancer Patient Cohort, CRCPC), age 40-74 years (CRC Screening Cohort, CRCSC)
* Newly-diagnosed colon and rectal cancer for stages Ⅰ-Ⅳ (CRCPC)

Exclusion Criteria:

* A history of colorectal cancer or bowel resection
* Non-Chinese speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NCRCC study consists of two subcohorts (CRC Screening Cohort and Colorectal Cancer Patient Cohort).
  CRC Screening Cohort is a population-bsaed study. All aged 40-74 years old individuals without prior colorectal cancer or bowel resection are recruited.
  All consecutive patients who were newly diagnosed with primary invasive or metastatic colorectal cancer are eligible for Colorectal Cancer Patient Cohort.
Sampling Method: Non-Probability Sample
Enrollment: 55000 (Estimated)
Dates: Start 2013-01-01 (Actual); Primary Completion 2035-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
colorectal cancer incidence | up to 15 years
Disease-free and overall survival | up to 10 years
Recurrence/metastasis | up to 5 years
Adenoma or advanced adenoma incidence | up to 1 year

SECONDARY OUTCOMES:
Prevalence of treatment-related toxicities characterized by the Common Toxicity Criteria for Adverse Events (CTCAE) | up to 5 years
Second primary cancer incidence | up to 15 years

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Second Affiliated Hospital Zhejiang University College of Medicine, Hangzhou, Zhejiang
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing
  - West China Hospital, Chengdu
  - Sun Yat-sen University, Guangzhou
  - Shanghai Zhongshan Hospital, Shanghai

REFERENCES:
- [Derived] Huang F, Xiao T, Li K, Wei R, Mei S, Zhao W, Wei F, He M, Zheng Z, Liu Q. Benefit of oxaliplatin-based chemotherapy or capecitabine monotherapy in older patients with stage III and high-risk stage II colon cancer: Data from the National Colorectal Cancer Cohort study in China. Chin Med J (Engl). 2025 Nov 10. doi: 10.1097/CM9.0000000000003813. Online ahead of print. PMID 41213862
- [Derived] Huang F, Jiang S, Wei R, Xiao T, Wei F, Zheng Z, Liu Q. Association of resection margin distance with anastomotic recurrence in stage I-III colon cancer: data from the National Colorectal Cancer Cohort (NCRCC) study in China. Int J Colorectal Dis. 2024 Jul 12;39(1):105. doi: 10.1007/s00384-024-04684-x. PMID 38995409